CLINICAL TRIAL: NCT00347802
Title: Diurnal Curves With Bimatoprost 0.03% Versus Travoprost 0.004%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 5176
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2007-06-01 (Estimated); Status verified 2007-05

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Bimatoprost

INTERVENTIONS:
Drug: Bimatoprost 0.03%, Travoprost 0.004%

SUMMARY:
To compare the diurnal curves in patients using bimatoprost 0.03% versus travoprost 0.004% for the treatment of glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* · Male or female > 18 years of age

  * Naive to treatment or washed off any ocular hypotensive agents
  * Untreated IOP >19 mm Hg
  * Diagnosis of open-angle glaucoma or ocular hypertension
  * Ability to provide informed consent and likely to complete study

Exclusion Criteria:

* · Known contraindication to bimatoprost or travoprost, or any component of any study medication

  * Uncontrolled systemic disease
  * Active ocular disease other than glaucoma or ocular hypertension
  * Required use of ocular medications other than the study medications during the study
  * History of intraocular surgery within the last 3 months
  * Prior discontinuation of any of the study medications for reasons related to efficacy or safety

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Robert Noecker, MD, Principal Investigator — UPMC Eye Center
Locations (1):
- Dr. Noecker, Pittsburgh, Pennsylvania, United States